CLINICAL TRIAL: NCT04336176
Title: Does a Novel Diabetic Foot Offloading Boot Reduce the Pressure Time Integral Compared to Usual Standard Care, in Patients With Diabetic Foot Ulcer? A Proof of Concept Pilot Study
Brief Title: Evaluating Plantar Foot Pressure in a Novel Diabetic Offloading Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Anne-Maree Keenan, Chair of Applied Health Research, University of Leeds
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 17/NS/0027
Record Dates: First submitted 2020-03-26; First posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Proof of concept study comparing the ability to redistribute forefoot pressure using a new foot offloading device compared to usual standard care. The sample will be purposively selected taken from a local population of active diabetic foot ulcer patients. The measurements will be taken from patients wearing usual standard of care, sham shoe (closest to barefoot or baseline pressures) and the PulseFlow DF boot. The measurements from each patient will be collated to compute pti averages for the comparison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PulseFlow DF boot (Active Comparator): PulseFlow DF boot
  Interventions: Device: PulseFlow DF boot; Device: Usual standard of care; Device: Sham
- Usual Care (Active Comparator): Measurements will be taken from patients wearing usual standard of care
  Interventions: Device: PulseFlow DF boot; Device: Usual standard of care; Device: Sham
- Sham (Sham Comparator): Sham shoe (closest to barefoot or baseline pressures)
  Interventions: Device: PulseFlow DF boot; Device: Usual standard of care; Device: Sham

INTERVENTIONS:
Device: PulseFlow DF boot — Offloading boot
Device: Usual standard of care — Usual standard of care (offloading device)
Device: Sham — Sham shoe (closest to barefoot or baseline pressures)

SUMMARY:
The impacts from diabetes are both patient related and healthcare based. Offloading is recognised as the priority treatment for healing neuropathic and neuro-ischaemic plantar foot ulcers. The new PulseFlow DF boot is a device which claims to off load but has little or no evidence on diabetic foot ulcer (DFU) subjects. Thus the primary aim of this study is to observe forefoot plantar pressures in a cross sectional purposively selected sample compared to usual standard of care.

DETAILED DESCRIPTION:
The impacts from diabetes are both patient related and healthcare based. DFU is associated with a high mortality rate at 34% at 1 year. There is an associated higher limb amputation rate from DFU than other causes. The high mortality rate, high amputation rate and increased socio-economic burden means providing high quality evidence based DFU service provision should be a NHS priority. Offloading is recognised as the priority treatment for healing neuropathic and neuro-ischaemic plantar foot ulcers. Since the provision of non removable devices or total contact casts (TCC) is poor, options have to be available that are equivalent in effectiveness at off loading and healing DFU. By improving the quality of offloading choices and acceptability for devices this will improve healing rates and reduce the cost burden where currently in the UK diabetic foot care in 2015 accounted for 0.6%/585.5million pounds of the NHS budget. The evidence for effectiveness of non removable devices is poor. Therefore any device that offloads to the equivalent or more than previous devices and current usual standard of care must be evidenced. The new PulseFlow DF boot is such a device which claims to off load but has little or no evidence on DFU subjects. Thus the primary aim of this study is to observe forefoot plantar pressures in a cross sectional purposively selected sample compared to usual standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Plantar forefoot diabetic foot ulcer over the 1st, 2nd, 3rd, 4th or 5th MTP joints
2. Neuropathic or Neuro-Ischaemic classification foot ulcer (taken from the TEXAS classification system)
3. Orthotic intervention for offloading/usual standard
4. English speaking and reading
5. Palpable foot pulses and/or Ankle Brachial Pressure Indices of values 0.8 to 1.29.

Exclusion Criteria:

1. Being treated for or having an active Charcot Arthropathy
2. Ankle Brachial Pressure Indices of <0.8 and >1.29. Using a standardised reproducible instrument called the Huntleigh Dopplex Ability Unit (DA100PB).
3. Purely ischaemic classification foot ulcer
4. Clinically active Infection causing lower leg swelling
5. Current active osteomyelitis
6. Due to alterations in gait, patients with diagnosed vascular dementia, Parkinson's, alcoholism or other major medically related gait alterations i.e. intoxication, brain cancers, muscular degeneration diseases, inflammatory arthritis, etc. This does not include osteo-arthritis.
7. Fractures of the foot
8. Pregnancy
9. Patients with forefoot trans metatarsal or major amputations
10. Temporary, accommodating or footwear not designed to offload used as their USC
11. Under another trial regarding foot dressings or off loading -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-07-29 (Actual)

PRIMARY OUTCOMES:
Pressure Time Integral | 1 day
  Gait analysis

SECONDARY OUTCOMES:
Modified Monitoring Orthopaedic Shoes questionnaire | 1 day (post gait analaysis)
  Multiple choice questionnaire and visual analogue pain scale measuring relevant factors of use and usability of orthopaedic shoes from a patient's perspective.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Maree Keenan, PhD, Study Chair — University of Leeds
Locations (1):
- The Leeds Teaching Hospitals NHS Trust., Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT04336176/Prot_SAP_000.pdf